CLINICAL TRIAL: NCT04050696
Title: The Safety and Efficacy of the Use of a Brain-computer Interface-based Electromagnetic Field Treatment in the Management of Chronic SCI Patients - a Pilot Study
Brief Title: The Use of Electromagnetic Field (EMF) Treatment in Chronic Spinal Cord Injury (SCI) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BrainQ Technologies Ltd. (Industry)
Collaborators: The Miami Project to Cure Paralysis (Other); Sheba Medical Center (Other Government); Kessler Institute for Rehabilitation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BQ4
Record Dates: First submitted 2019-07-30; First posted 2019-08-08 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Incomplete Spinal Cord Injury
Keywords: chronic SCI; incomplete SCI; central cord syndrome; electromagnetic field; physical therapy; cervical SCI; paraplegia; tetraplegia; upper limb impairment; GRASSP; ISNCSCI
MeSH Terms: conditions — Central Cord Syndrome; Paraplegia; Quadriplegia

STUDY DESIGN:
Masking Description: Treatment-only study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment (with PT run-in) (Experimental): Treatment group, to receive BQ treatment with PT, after stability established in 4 week PT run-in period
  Interventions: Device: BQ 1.2

INTERVENTIONS:
Device: BQ 1.2 — BQ 1.2 exposure of EMF exposure paradigm in conjunction with upper limb PT regimen

SUMMARY:
The purpose of this study is to further establish safety and efficacy of the BQ EMF treatment of chronic SCI subjects who demonstrate stability in The Graded and Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) strength score following a one-month physical therapy run-in period.

DETAILED DESCRIPTION:
BQ is a brain-computer interface (BCI) based medical device that produces and delivers non-invasive, low intensity and low frequency electromagnetic fields targeting a patient's central nervous system (CNS) for motor rehabilitation. The technology behind the device utilizes machine learning (ML) tools to identify high-resolution spectral patterns, which characterize motor functions within EEG and MEG/EMG measurements taken during functional motor tasks. These patterns are then translated into a frequency-dependent, low intensity and non-invasive electromagnetic treatment, which applies similar patterns directly to a patient's CNS.

BQ treatment is intended to improve upper limb motor function of chronic SCI patients, over 18 years of age with an incomplete injury and upper limb motor impairment (AIS B - D, Cervical C1 - C8). The treatment will be administered as an adjunctive treatment along with a typical pharmacological and/or non-pharmacological treatment plan.

Study is a prospective, single arm, multicenter study with physical therapy (PT) run-in phase, where each subject serves as his/her own control. Study population will include at least 8 individuals with traumatic or (incident-related) non-traumatic chronic cervical incomplete SCI (AIS B-D) who are 12 - 30 months post-injury, with score between 5 - 35 on GRASSP strength subscore on at least one side, and medically stable.

The primary objective of this study is to evaluate the efficacy of the BQ system treatment in improving upper limb motor function of chronic SCI subjects, compared to their own baseline after stability has been demonstrated during physical therapy run-in period, as measured by improvement in GRASSP strength subscore. An additional secondary objective of the study is to evaluate the efficacy of the BQ system treatment in improving motor recovery, spasticity, pain, QOL, and imaging outcomes in the stated population.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females who are between 18 to 75 years of age
2. Diagnosed with traumatic or (incident-related) non-traumatic chronic cervical incomplete SCI (AIS B-D), 12 to 30 months from event.
3. Individuals with a score between 5 - 35 on the GRASSP strength subscore on at least one side
4. Medically stable
5. Cognitive status and ability to communicate must be at a level consistent with that which is required to participate in motor rehabilitation regimen (e.g. can follow directions and cued tasks)
6. Stable pharmacological treatment plan without any planned modifications
7. Able to engage in physical therapy program as stipulated per protocol
8. Passive shoulder flexion of at least 60 degrees and passive shoulder abduction of at least 40 degrees, to ensure ability to perform upper limb motor tasks
9. Negative pregnancy test in women of childbearing potential
10. Subject can independently provide consent (written or verbal in the presence of a family member) to participate in the study and is willing to comply with study procedures

Exclusion Criteria:

Subjects not eligible for this study include those that have any of the following:

1. Excessive pain in the UE that limits the administration of the evaluation measurements
2. Excessive spasticity: subjects with MAS of wrist ≥ 2, or MAS of elbow ≥ 3
3. Received botulinum toxin in the previous 4 months, or planning of an upcoming injection during the trial period
4. Participating in any other experimental rehabilitation or drug studies
5. Medical conditions or circumstances that, in the opinion of the investigators, would preclude safe and/or effective participation
6. Severe cognitive or psychiatric problems that might significantly impact the successful study conduct
7. History of epileptic seizures or epilepsy
8. Implanted electronic medical devices
9. Alcoholism or drug addiction as defined by DSM-IV within last 5 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of treatment to end of treatment in the Graded and Redefined Assessment of Strength, Sensibility and Prehension (GRASSP - strength subscore): | Week 22
  The GRASSP is a clinical measure of upper limb impairment, which incorporates the construct of upper limb sensorimotor function. This measurement captures information on upper limb sensorimotor impairment for individuals with tetraplegia and defines neurological status with numerical values, which represent the deficits in a predictive pattern. The GRASSP demonstrates reliability, construct validity, and concurrent validity for use as a standardized upper limb impairment measure for individuals with incomplete SCI (Kalsi-Ryan et al., 2012). Scores can be used to determine relationships between impairment and functional capability of the upper limb.
  The evaluation includes three domains of hand function:
  1. Strength (primary)
  2. Sensibility (secondary)
  3. Prehension (secondary)
  For the primary outcome measure, only the strength subscore will be assessed as follows:
  ● Strength (10 muscles of arm & hand): motor grade 0-5 for each (sum = subtest total, 0-50)

SECONDARY OUTCOMES:
GRASSP (strength subscores) | Week -1, week 1, week 5, week 9, week 14, week 18, week 22, week 26, week 34
  The GRASSP is a clinical measure of upper limb impairment, which incorporates the construct of upper limb sensorimotor function. This measurement captures information on upper limb sensorimotor impairment for individuals with tetraplegia and defines neurological status with numerical values, which represent the deficits in a predictive pattern. The GRASSP demonstrates reliability, construct validity, and concurrent validity for use as a standardized upper limb impairment measure for individuals with incomplete SCI (Kalsi-Ryan et al., 2012). Scores can be used to determine relationships between impairment and functional capability of the upper limb.
  ● Strength (10 muscles of arm & hand): motor grade 0-5 for each (sum = subtest total, 0-50)
GRASSP (sensibility and prehension subscores) | Week -1, week 1, week 5, week 9, week 14, week 18, week 22, week 26, week 34
  For the secondary outcome measure, the sensibility and prehension subscores will be assessed as follows:
  * Dorsal sensation (3 locations): each scored 0-4 (sum = subtest score, 0-12)
  * Palmar sensation (3 locations): each scored 0-4 (sum = subtest score, 0-12)
  * Prehension ability: 3 grasps (cylindrical, lateral key, tip to tip), each scored 0-4 (sum = 0-12).
  * Prehension performance: 6 prehension tasks - pour water from bottle, pick up an object, transfer 9 pegs from board to board, screw four nuts onto bolts, each scored 0-5 (sum = subtest score, 0-30).
ISNCSCI (International Standards for Neurological Classification of Spinal Cord Injury) | Week -1, week 1, week 5, week 9, week 14, week 18, week 22, week 26, week 34
  This is a system of tests used to define and describe the extent and severity of a subject's spinal cord injury. The subject's grade is based on how much sensation he or she can feel at multiple points on the body, as well as tests of motor function.
  For the purposes of this study, only the motor subtests and functions (UEMS & LEMS) will be considered as a secondary outcome measure.
  The full ISNCSCI will be administered and assessed at baseline and end of treatment only for AIS classification purposes.
Modified Ashworth Scale (MAS) | Week -1, week 1, week 5, week 22
  The Modified Ashworth scale (MAS) measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity (Bohannon & Smith, 1987). Scoring are as follows:
  * 0: No increase in muscle tone
  * 1: Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  * 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  * 2: More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  * 3: Considerable increase in muscle tone, passive movement difficult
  * 4: Affected part(s) rigid in flexion or extension
Spinal Cord Independence Measure III (SCIM III - self-care sub-score) | Week 1, week 5, week 9, week 14, week 18, week 22, week 26, week 34
  The Spinal Cord Independence Measure (SCIM) is a disability profile containing 3 sub-scales developed specifically for people with spinal cord injury (SCI). Through measures across its distinct scales, the profile describes subjects' ability to undertake activities of daily living (Ackerman, Morrison, McDowell, & Vazquez, 2010). Each area is scored according to its proportional weight in these subjects' general activity. The final score ranges from 0 to 100 (Ackerman et al., 2010). The SCIM includes the following areas of function:
  * Self-care (sub-score 0 - 20)
  * Respiration and sphincter management (sub-score 0 - 40)
  * Mobility (sub-score 0 - 40)
Questionnaire of von Korff et al. Grading the Severity of Chronic Pain | Week 1, week 5, week 22
  This is a simple method of grading the severity of chronic pain. This questionnaire grades the severity of chronic pain based on its characteristics and its impact on a person's activities (Von Korff, Ormel, Keefe, & Dworkin, 1992).
  Answers are graded on a 0 (no) - 10 (extreme) scale for each of the following questions:
  * Rate pain at present time
  * Rate of most intense pain in the last 6 months
  * Rate of average pain in the last 6 months
  * In the past 6 months, how has pain interfered with your daily activities
  * In the past 6 months, how has pain interfered with your recreational social and family activities
  * In the past 6 months, how has pain interfered with your ability to work
Capabilities of the Upper Extremity Test (CUE-T) | Week 1, week 5, week 22
  A 32-item questionnaire with items in seven domains. The CUE test displays excellent test/retest reliability, and excellent correlation with impairment and capacity measures in persons with incomplete SCI. Subjects are scored on a 7-point scale representing self-perceived difficulty: 1 indicating totally limited, can't do at all, and 7 indicating not at all limited. Minimum score is 32 and maximum score is 124 (Marino, Shea, & Stineman, 1998).
  Subjects will be asked to complete the following tasks:
  * 15 unilateral (left and right) items
  * 2 bilateral items
  * 3 reaching items
  * 4 pulling/pushing items
  * 2 wrist items
  * 6 hand/finger items
  * 2 bilateral items
The Spinal Cord Injury-Quality of Life (SCI-QOL) | Week 1, week 5, week 22
  The measurement system was developed to address the shortage and non-uniformity of subject-reported outcome measures for clinical care and research in SCI rehabilitation. It consists of 19 items, measuring emotional health (depression, anxiety, resilience, positive affect and well-being, grief/loss, self-esteem, stigma, psychological trauma); physical-medical health (bowel management, bladder management, bladder complications, pressure ulcers, pain interference, pain behavior); social participation (ability to participate in social roles and activities, satisfaction with social roles and activities, independence); physical function (basic mobility, self-care, fine motor functioning, wheelchair mobility, ambulation) (Tulsky et al., 2015).
Magnetic Resonance Imaging (MRI) and Diffusion Tensor Imaging (DTI) scans | Week 5, week 22
  For applicable subjects, MRI scans will be performed, preferably with a 3.0 T Ingenia Philips scanner, according to the follow sequences:
  A. Sagittal T2 B. Sagittal STIR C. Sagittal PW (proton density) D. Sagittal T1 E. Sagittal DTI F. Axial T1 G. Axial T2 MRI results will be analyzed to quantify tissue integrity (e.g. white matter, grey matter, cerebrospinal fluid). DTI measurements will be used to identify water movement, which, in the CNS, is often localized within axons, and provides high contrast towards white matter, indicating the quality and quantity of nerve fibers. This endpoint is not obligatory per protocol; failure to complete in contraindicated subjects is not considered a protocol deviation per Good Clinical Practice.

OTHER OUTCOMES:
Surface EEG | Week 1, week 5, week 9, week 14, week 18, week 22, week 26
  Surface EEG will be recorded throughout the trial to gauge subject progress. This endpoint is exploratory, and will not be used for diagnostic or inclusionary/exclusionary purposes.
Surface EMG | Week 1, week 5, week 9, week 14, week 18, week 22, week 26
  Surface EMG will be recorded throughout the trial to gauge subject progress. EMG will be recorded in a bipolar setting from electrode pairs on the following muscles: flexor carpi radialis brevis, extensor carpi radialis brevis, flexor carpi ulnaris, extensor carpi ulnaris. The subjects will be seated and requested to perform hand and arm movements, to their best ability, upon cues. This endpoint is exploratory, and will not be used for diagnostic or inclusionary/exclusionary purposes.
Smoothness of reaching movement | Week 1, week 5, week 9, week 14, week 18, week 22, week 26, week 34
  Upper extremity (UE) kinematics data will be collected using a motion capture system. Retro-reflective markers will be attached directly to the subject with use of double sided tape on the anatomical joint mark points using the modified Helen Hayes marker set (torso, head and upper extremity). All kinematic data will be collected and time matched with the EMG data and transferred to a custom MATLAB (Mathworks, Natick, MA) algorithm code for further analysis.
  Upper extremity joint kinematics, muscle activation (sEMG) and EEG data will be recorded during several activities.
  To evaluate the smoothness of movements, the third derivative of the UE joint angles will be computed and considered for estimation of smoothness at the shoulder, elbow and wrist joints.
Range of motion (ROM) | Week 1, week 5, week 9, week 14, week 18, week 22, week 26, week 34
  Upper extremity (UE) ROM (in the sagittal, frontal, and transverse planes) will be collected using a motion capture system. Retro-reflective markers will be attached directly to the subject with use of double sided tape on the anatomical joint mark points using the modified Helen Hayes marker set (torso, head and upper extremity).
  Upper extremity ROM, muscle activation (sEMG) and EEG data will be recorded during several activities.
Venous blood collection | Week 1, week 5, week 22
  Five ml whole venous blood will be collected at baseline (W5), midterm (W14), at end of treatment phase (W22), and first follow-up (W26) from all subjects. Blood will be separated to two test tubes, 2.5 CC in each, one with anti-coagulant (EDTA) and one without. Red blood cells will be separated from plasma (EDTA tube, by centrifugation) or from serum by clotting. Plasma and serum samples will be frozen in 0.5 cc aliquots at -80°C. Samples will be analyzed for CNS insult biomarkers, including glial fibrillary acidic protein (GFAP) and ubiquitin carboxy-terminal hydrolase L1 (UCH-L1), as well as brain-derived neurotrophic factor (BDNF), vascular endothelial growth factor (VEGF), and nerve growth factor beta (NGFβ). This draw is an exploratory endpoint, and is not obligatory PP if contraindicated.
Assessment of device's Usability by user (Human factors and usability analysis) | Week 0 of 1st patient, week 22 of 2nd patient, week 34 of 4th patient
  Usability form to be completed by device user (operator) shall include:
  1. Subjective feedback questionnaire: Subjective feedback focusing on any concerns on using device, ease of use, and potential deviations from proper use.
  2. Informative questions to ensure proper understanding and operation of the device.
  The form is designed in order to track possible deviations from required treatment due to human factors, as well as specific elements of the treatment which may pose a risk due to human factors and have not been accounted for in the design and validation process.
Rate of deviation of device user from expected input sequence (Human factors and usability analysis) | Week 34 of 4th patient
  Deviation of device user from expected input sequence, defined as exiting the "treatment flow" during treatment or canceling treatment unnecessarily, and obtained by user activity logging. The expectation is that these deviations should occur in less than 10% of treatment sessions

CONTACTS AND LOCATIONS:
Overall Officials: Gabi Zeilig, Ph.D., Principal Investigator — Sheba Medical Center; Dalton Dietrich, Ph.D., Principal Investigator — The Miami Project to Cure Paralysis; Ghaith Androwis, Ph.D., Principal Investigator — Kessler Institute of Rehabilitation
Locations (3):
- United States (2):
  - The Miami Project to Cure Paralysis, Miami, Florida
  - Kessler Institute of Rehabilitation, West Orange, New Jersey
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No
Metadata can be made available, upon reasonable request Individual patient data (IPD) to be shared if significant need/benefit can be demonstrated, and only with permission of individual subject, as it is not specifically covered in informed consent form (ICF)